CLINICAL TRIAL: NCT04406779
Title: The Frequency of Thyroid Diseases in Women With Breast Cancer
Status: Completed | Type: Observational
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Cevdet Duran, M.D., Uşak University
Other Study IDs: UsakU-Cevdet1
Record Dates: First submitted 2020-05-22; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Breast Cancer; Thyroid Diseases
MeSH Terms: conditions — Breast Neoplasms; Thyroid Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with breast cancer: Patients with breast cancer
  Interventions: Device: thyroid USG was perform, blood samples were taken for the meausurement of thyroid hormone and autoantibodies
- Control: Healthy patients without breast cancer
  Interventions: Device: thyroid USG was perform, blood samples were taken for the meausurement of thyroid hormone and autoantibodies

INTERVENTIONS:
Device: thyroid USG was perform, blood samples were taken for the meausurement of thyroid hormone and autoantibodies — thyroid USG was perform, blood samples were taken for the meausurement of thyroid hormone and autoantibodies

SUMMARY:
Breast cancer and thyroid disorders are important health challenges commonly encountered in women. The relationship between both conditions still remains unknown. In this study, the frequency of thyroid diseases was investigated in breast cancer patients

ELIGIBILITY:
Inclusion Criteria:

* women, the age between 18-65 years who were diagnosed with breast cancer, but not underwent surgery, radiotherapy or chemothreapy were included into the study

Exclusion Criteria:

* Those with pregnancy, known liver and renal failure, the history of any malignancy other than breast cancer, undergoing a surgical operation due to breast cancer, also those receiving chemotherapy/radiotherapy for the same reason or undergoing partial or complete thyroid surgery or a surgical operation within the past 6 months, and also the patients taking oral anti-diabetic medication, insulin, steroids, thiazide, anti-psychotics and immuno-suppressive medicines affecting the levels of blood glucose, insulin and IR, smokers and those consuming alcohol were excluded

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: women, aged between 18-65 years who were diagnosed with breast cancer, but not underwent surgery, radiotherapy or chemothreapy were included into the study as patients groups. Age matched healthy controls were enrolled as controls.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
to investigate the frequency of thyroid diseases in breast cancer patients. | 1 year

IPD SHARING:
Plan to Share IPD: No